CLINICAL TRIAL: NCT05356897
Title: 3T: a Phase II Single Arm Open Label Study of Tucatinib Combined with Trastuzumab and TAS-102 in Molecularly Selected Patients with HER2+ Metastatic Colorectal Cancer
Brief Title: Tucatinib Combined with Trastuzumab and TAS-102 for the Treatment of HER2 Positive Metastatic Colorectal Cancer in Molecularly Selected Patients, 3T Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no sites were regulatory ready and the SC took the study to a different group.
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-GI-2003; NCI-2022-03147 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-GI-2003 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Colon Adenocarcinoma; Metastatic Colorectal Adenocarcinoma; Metastatic Rectal Adenocarcinoma; Stage IV Colon Cancer AJCC V8; Stage IV Colorectal Cancer AJCC V8; Stage IV Rectal Cancer AJCC V8
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — Trastuzumab; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02; Trifluridine; trifluridine tipiracil drug combination; tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (tucatinib, trastuzumab, TAS-102) (Experimental): Patients receive tucatinib PO BID, trastuzumab IV over 30-90 minutes on days 1 and 15, and TAS-102 PO BID on days 1-5 and 8-12. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Trastuzumab; Drug: Trifluridine and Tipiracil Hydrochloride; Drug: Tucatinib

INTERVENTIONS:
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herzuma; Kanjinti; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; Ontruzant; PF-05280014; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-pkrb; Trastuzumab-qyyp; Trazimera
Drug: Trifluridine and Tipiracil Hydrochloride — Given PO
  Other Names: Lonsurf; TAS 102; TAS-102; Tipiracil Hydrochloride Mixture with Trifluridine; Trifluridine/Tipiracil; Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102
Drug: Tucatinib — Given PO
  Other Names: ARRY-380; Irbinitinib; ONT-380; Tukysa

SUMMARY:
This phase II trial studies whether tucatinib combined with trastuzumab and TAS-102 works to shrink tumors in patients with HER2 positive colorectal cancer that has spread to other parts of the body (metastatic) and has one of the following gene mutations detected in blood: PIK3CA, KRAS, NRAS, or BRAF V600. Tucatinib is in a class of medications called kinase inhibitors. It works by blocking the action of the abnormal protein that signals tumor cells to multiply. This helps stop or slow the spread of tumor cells. Trastuzumab is a form of targeted therapy because it attaches itself to specific molecules (receptors) on the surface of tumor cells, known as HER2 receptors. When trastuzumab attaches to HER2 receptors, the signals that tell the cells to grow are blocked and the tumor cell may be marked for destruction by the body's immune system. TAS-102 is a combination of 2 drugs; trifluridine and tipiracil. Trifluridine is in a class of medications called thymidine-based nucleoside analogues. It works by stopping the growth of tumor cells. Tipiracil is in a class of medications called thymidine phosphorylase inhibitors. It works by slowing the breakdown of trifluridine by the body. Giving tucatinib, trastuzumab, and TAS-102 together may work better than usual treatment for metastatic colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the 2-month progression free survival (PFS) rate of tucatinib, trastuzumab, and trifluridine and tipiracil hydrochloride (TAS-102) in patients with HER2 amplified and PIK3CA, RAS, and/or BRAF mutated metastatic colorectal cancer (CRC).

SECONDARY OBJECTIVES:

I. To assess the clinical benefit rate (CBR) (stable disease [SD] for >= 4 months, or best response of complete response [CR] or partial response [PR]) of tucatinib, trastuzumab, and TAS-102 in patients with HER2 amplified and PIK3CA, RAS, and/or BRAF mutated metastatic CRC.

II. To assess the objective response rate (ORR) of tucatinib, trastuzumab, and TAS-102 in patients with HER2 amplified and PIK3CA, RAS, and/or BRAF mutated metastatic CRC.

III. To assess the overall survival (OS) of tucatinib, trastuzumab, and TAS-102 in patients with HER2 amplified and PIK3CA, RAS, and/or BRAF mutated metastatic CRC.

IV. To assess the safety and tolerability of tucatinib, trastuzumab, and TAS-102 in patients with HER2 amplified and PIK3CA, RAS, and/or BRAF mutated metastatic CRC.

CORRELATIVE RESEARCH OBJECTIVES:

I. To assess whether the combination of tucatinib, trastuzumab, and TAS-102 eliminates HER2 amplified circulating tumor deoxyribonucleic acid (DNA) (ctDNA) from peripheral blood.

II. To explore the correlation between tissue and blood-based biomarkers and clinical outcomes.

OUTLINE:

Patients receive tucatinib orally (PO) twice daily (BID), trastuzumab intravenously (IV) over 30-90 minutes on days 1 and 15, and TAS-102 PO BID on days 1-5 and 8-12. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days and then every 12 weeks for 4 years after study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Registered to COLOMATE ACCRU-GI-1611 and:

  * COLOMATE Companion Trial Recommendation Form indicates patient meets molecular eligibility for enrollment to this study (at least one of the following: PIK3CA, KRAS, NRAS, or BRAF V600 mutation detected in blood from the Guardant360 assay)
  * COLOMATE Companion Trial Recommendation Form date of completion is < 90 days prior to registration
* Age >= 18 years
* Histologically and/or cytologically confirmed metastatic adenocarcinoma of the colon or rectum
* Life expectancy >= 3 months in the estimation of the investigator
* Previous treatment with or contraindication to:

  * A fluoropyrimidine (e.g., 5-fluorouracil or capecitabine)
  * Oxaliplatin
  * Irinotecan
  * An anti-VEGF biological therapy (including but not limited to bevacizumab, ramucirumab, or ziv-aflibercept)
  * If the tumor has deficient mismatch repair proteins or is microsatellite instability (MSI)-High based on tumor tissue testing, an anti-PD-1 monoclonal antibody (nivolumab or pembrolizumab)
  * (Cancer Therapy List [colorectal cancer] is available on the Academic and Community Cancer Research United [ACCRU] web site)
* Radiographically measurable disease as per Response Evaulation Criteria in Solid Tumors (RECIST) version 1.1
* Molecular testing result from Clinical Laboratory Improvement Act (CLIA)-certified laboratory confirming that the tumor tissue has at least one of the following:

  * HER2 3+ by immunohistochemistry (IHC)
  * HER2 2+ by IHC and HER2 (ERBB2) amplification by in situ hybridization assay (Signal ratio > 2.2 or gene copy number > 6 by either fluorescence in situ hybridization (FISH) or chromogenic in situ hybridization (CISH)
  * HER2 (ERBB2) amplification by CLIA-certified next generation sequencing (NGS) assay
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1, or 2 (Form is available on the ACCRU web site)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 7 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 7 days prior to registration)
* Hemoglobin > 8.0 g/dL (obtained =< 7 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 7 days prior to registration)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 3 X upper limit of normal (ULN) (obtained =< 7 days prior to registration)
* Creatinine clearance (using Cockcroft and Gault equation) >= 50 mL/min or serum creatinine less than 1.5 x the upper limit of institutional normal (ULN) (obtained =< 7 days prior to registration)
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless on medication known to alter INR and/or aPTT (obtained =< 7 days prior to registration)
* Negative serum pregnancy test =< 7 days prior to registration for women of childbearing potential only. Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Post menopause is defined as amenorrhea >= 12 consecutive months Note: Women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, ovarian suppression or any other reversible treatment
* Sexually active subjects (men and women) agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used
* Willing to provide informed written consent =< 30 days prior to registration
* Left ventricular ejection fraction (LVEF) >= 50% as assessed by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA) documented =< 28 days prior to registration
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).

  * Note: During the Active Monitoring Phase of a study (i.e., active treatment and clinical follow-up), participants must be willing to return to the consenting institution for follow-up
* Willing to provide tissue and blood samples for correlative research purposes
* Willing to allow transfer of tissue and blood samples, clinical information, and outcome data collected from this trial for future research

Exclusion Criteria:

* Radiation therapy, hormonal therapy, biologic therapy, experimental therapy, or chemotherapy for cancer < 21 days prior to registration
* Prior treatment with an anti-HER2 tyrosine kinase inhibitor, including but not limited to tucatinib, lapatinib, or neratinib

  * Note: Prior treatment with an anti-HER2 antibody or antibody drug conjugate is permitted (including but not limited to trastuzumab, pertuzumab, fam-trastuzumab-deruxtecan-nxki, ado-trastuzumab emtansine)
* Prior treatment with TAS-102
* Concurrent severe and/or uncontrolled medical conditions which may compromise participation in the study, including impaired heart function or clinically significant heart disease
* Not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 =< Grade 1 from toxicity due to all prior therapies except alopecia, oxaliplatin-related neuropathy, and clinically insignificant electrolyte abnormalities. Congestive heart failure (CHF) must have been =< Grade 1 in severity at the time of occurrence and must have resolved completely prior to registration
* Female patients who are pregnant or breast feeding
* Currently taking medications specified by the protocol as prohibited for administration in combination with study drug
* Known active central nervous system (CNS) metastases (patients with radiated or resected lesions are permitted, provided the lesions are fully treated and inactive, patients are asymptomatic, and no steroids have been administered >= 30 days prior to registration)

  * Note: Steroids for treatment of other medical conditions other than CNS metastases are permitted
* Inability to swallow pills or any significant gastrointestinal disease which would preclude the adequate oral absorption of medications
* Use of a strong cytochrome P450 (CYP)2C8 inhibitor within 5 half-lives of the inhibitor or use of a strong CYP3A4 or CYP2C8 inducer within 5 days prior to registration
* Major surgical procedure, open biopsy, or significant traumatic injury =< 28 days prior to registration (56 days for hepatectomy, open thoracotomy, major neurosurgery) or anticipation of need for major surgical procedure during the course of the study
* Serious, non-healing wound, ulcer, or bone fracture
* History of stroke (cerebrovascular accident), transient ischemic attack (TIA), myocardial infarction (MI), unstable angina, cardiac or other vascular stenting, angioplasty, or cardiac surgery =< 6 months prior to registration
* Known history of congestive heart failure - New York Heart Association (NYHA) >= Class II (See NYHA Classifications on the ACCRU website)
* Known history of human immunodeficiency virus (HIV) seropositivity, acute or chronic active hepatitis B or C infection, or other serious chronic infection requiring ongoing treatment
* Known chronic liver disease, autoimmune hepatitis, or sclerosing cholangitis
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Any previously untreated or concurrent cancer that is distinct in primary site or histology from colorectal cancer except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor.

  * Note: Subjects surviving a cancer that was curatively treated and without evidence of disease or biochemical relapse (undetectable prostate-specific antigen [PSA] for prostate cancer) for 3 or more years before registration are allowed. All cancer treatments must be completed at least 3 years prior to registration
* Unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate | At 2 months
  Defined as progression-free and alive at the 2 months disease evaluation scan. Disease status will be assessed using Response Evaluation Critera in Solid Tumors (RECIST) version (v). 1.1. Evaluable patients are defined as those who are eligible, consented, and received any protocol treatment. A 95% confidence interval will be calculated using the method proposed by Koyama and Chen, 2008 and implemented with the R software package clinfun (RStudio, 2021; Venkatraman, 2018).

SECONDARY OUTCOMES:
Clinical benefit | Up to 4 years
  Defined as achieving complete response (CR), partial response (PR), or stable disease (SD) for at least 4 months while on treatment. Disease status will be assessed using RECIST v. 1.1 criteria. Clinical Benefit Rate will be calculated as the proportion of evaluable patients who achieve clinical benefit. The final CBR point estimate and corresponding 95% confidence interval calculated using the binomial exact method (Clopper & Pearson, 1934).
Overall response | Up to 4 years
  Defined as achieving CR or PR while on treatment. Disease status will be assessed using RECIST v. 1.1 criteria. Overall Response Rate will be calculated as the proportion of evaluable patients who achieve response. The final ORR point estimate and corresponding 95% confidence interval calculated using the binomial exact method.
Overall survival (OS) | From registration to death from any cause, assessed up to 4 years
  Will be estimated using the Kaplan-Meier method. Patients who are alive will be censored at the last follow-up date. The report will include the median OS and corresponding 95% confidence interval, which will be calculated using the method proposed by Brookmeyer and Crowley, 1982.
Incidence of adverse events | Up to 4 years
  All patients who have initiated treatment will be considered evaluable for adverse event analyses. The rate of patients experiencing a grade 3+ adverse event will be reported. Further analyses of adverse event rates will be considered exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: John H Strickler, Principal Investigator — Academic and Community Cancer Research United
Locations (2):
- United States (2):
  - UC San Diego Moores Cancer Center, San Diego, California
  - Duke University Medical Center, Durham, North Carolina